CLINICAL TRIAL: NCT00967954
Title: A Study of Changes in the Prostate Following Androgen Deprivation to Investigate Therapy Response and Resistance in Clinical Prostate Cancer
Brief Title: Study of Blood and Tissue Samples From Patients Receiving Androgen Deprivation for Newly Diagnosed Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: CDR0000639017; CRUK-CHIRRP; EU-20920
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2009-08

CONDITIONS: Prostate Cancer
Keywords: stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists; Comparative Genomic Hybridization; Gene Expression Profiling; Magnetic Resonance Spectroscopy

INTERVENTIONS:
Drug: antiandrogen therapy
Drug: releasing hormone agonist therapy
Genetic: DNA analysis
Genetic: RNA analysis
Genetic: comparative genomic hybridization
Genetic: gene expression analysis
Other: laboratory biomarker analysis
Procedure: diffusion-weighted magnetic resonance imaging
Procedure: magnetic resonance spectroscopic imaging

SUMMARY:
RATIONALE: Studying samples of blood and tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research study is looking at blood and tissue samples from patients with prostate cancer receiving androgen deprivation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify the molecular and pathophysiological changes which occur during the early stages of androgen deprivation (AD) and during emerging castration-resistant prostate cancer.
* To test functional imaging as a non-invasive tool to measure treatment response and validate this using biological endpoints.
* To develop clinical models to predict how tumors will respond to AD and identify new targets once AD fails.

OUTLINE:

* Group A: Patients likely to receive androgen deprivation (AD) as first-line therapy undergo blood and prostate biopsy sample collection before and after treatment on days 0 and 14 or 90. Patients receive an androgen receptor inhibitor followed by maintenance with a gonadotropin-releasing hormone analogue beginning on day 0. Patients also undergo diffusion-weighted MRI, MR spectroscopic imagining, quantitative T1W mapping, and T1W perfusion sequence.
* Group B: Patients already receiving AD undergo blood and prostate biopsy sample collection within 4 weeks of diagnosis of castration-resistant prostate cancer and before initiating any second-line therapy.

Blood and tissue samples are assessed via DNA and RNA genetic analysis, gene expression studies, and comparative genomic hybridization to identify novel markers of androgen response and resistance.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * High clinical suspicion of prostate cancer, based on an abnormal digital rectal examination and PSA (> 20 ng/mL)
  * Newly diagnosed, castration-resistant prostate cancer

    * Clinical stage ≥ T2c disease
* Significant tumor volume on initial diagnostic biopsy (> 50% of cores)
* Likely to receive androgen deprivation therapy for prostate cancer

PATIENT CHARACTERISTICS:

* No contraindication to transrectal needle biopsy
* No contraindication to MRI or prostate needle biopsy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-09; Primary Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Identification of molecular and pathophysiological changes
Functional imaging as a non-invasive tool to measure treatment response
Development of clinical models to predict tumor response

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Gnanapragasam, MD, Principal Investigator — Cancer Research UK
Locations (1):
- Cancer Research UK at Cambridge Research Institute, Cambridge, England, United Kingdom